CLINICAL TRIAL: NCT02597790
Title: Clinical and Translational Science Institute Prospective Longitudinal Assessment of Coinfected Subjects With HIV/Hepatitis C for Endothelial Function Study
Brief Title: A Prospective, Longitudinal Study of Endothelial Function in HIV/HCV Coinfected Subjects
Acronym: CTSI-PLACE
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kara Chew, Assistant Clinical Professor, University of California, Los Angeles
Other Study IDs: 12-001792 (CTSI-PLACE); N/A (Parent P30AI028697) (Other Grant/Funding Number: UCLA AIDS Institute/Center for AIDS Research); N/A (Parent UL1TR000124) (Other Grant/Funding Number: UCLA Clinical and Translational Science Institute); 52767 (Other Grant/Funding Number: Merck Investigator Studies Program)
Record Dates: First submitted 2015-10-30; First posted 2015-11-05 (Estimated); Results first posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-12

CONDITIONS: HIV; Hepatitis C
Keywords: endothelial function; cardiovascular risk; HIV; Hepatitis C; metabolic disease; inflammation
MeSH Terms: conditions — Hepatitis C; Metabolic Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A (HIV/HCV coinfected)
- Group B (HIV monoinfected)

SUMMARY:
The CTSI-PLACE Study is a study for men and women with HIV/hepatitis C co-infection or HIV only. The study looks at the impact of having hepatitis C virus in addition to HIV on risk for cardiovascular disease. Participants will undergo non-invasive assessment of cardiovascular disease risk through measurements of endothelial function and blood biomarkers at baseline and 1 year (or 4 weeks and 24 weeks after end of HCV treatment for those that undergo HCV treatment during study follow-up).

ELIGIBILITY:
Inclusion Criteria

1. Men and women ≥ 18 years
2. Hepatitis C negative or chronic hepatitis C infection
3. Chronic HIV infection
4. CD4+ T-cell count > 200 cells/mm3
5. Plasma HIV-1 RNA < 50 copies/mL
6. On continuous and stable ART for at least 12 weeks
7. Ability and willingness to provide written informed consent.

Exclusion Criteria

1. Known cardiovascular disease
2. Diabetes requiring insulin therapy or hemoglobin A1c > 8%
3. Inability to conform to requirements for PAT testing
4. Decompensated liver disease
5. Other known causes of significant liver disease
6. Serious illness including acute liver-related disease and malignancy requiring systemic treatment or hospitalization within 12 weeks prior to study entry
7. Presence of active or acute AIDS-defining opportunistic infections (OIs) within 12 weeks prior to study entry
8. History of major organ transplantation with an existing functional graft and on immunosuppressive therapy
9. History of known vascular or autoimmune disease
10. Pregnancy
11. HCV treatment (any approved or investigational agents) within 24 weeks prior to study entry
12. Use of immune-based therapies or systemic corticosteroids within 12 weeks prior to study entry
13. Advanced renal insufficiency as defined by glomerular filtration rate (GFR) < 30 mL/min/1.73 m2 or treatment by dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV/HCV coinfected and HIV monoinfected adults with well-controlled HIV
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2013-10; Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara W. Chew, M.D., M.S., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA CARE Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (HIV/HCV Coinfected): HIV+, HCV viremic at study entry
- Group B (HIV Monoinfected): HIV+, HCV negative at study entry
Period: Overall Study
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Started | 45 | 41
Completed | 36 | 29
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected) | Total
Number analyzed (Participants) | 45 | 41 | 86
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [46 to 57] | 52 [46 to 55] | 52 [46 to 55]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Men | 38 | 35 | 73
  Gender: Women | 4 | 4 | 8
  Gender: Transgender women | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black Non-Hispanic | 17 | 10 | 27
  Race/Ethnicity: White Non-Hispanic | 9 | 8 | 17
  Race/Ethnicity: Hispanic | 17 | 20 | 37
  Race/Ethnicity: Other | 2 | 3 | 5
Body mass index (kg/m2) [Median (Inter-Quartile Range); unit: kg/m2] | 27.6 [23.5 to 29.8] | 26.0 [23.7 to 27.5] | 26.3 [23.5 to 28.6]
Hypertension [Count of Participants; unit: Participants] | 11 | 7 | 18
Dyslipidemia [Count of Participants; unit: Participants] | 7 | 25 | 32
CD4+ T cell count [Median (Inter-Quartile Range); unit: cells/mm3] | 587 [405 to 794] | 636 [472 to 897] | 612 [445 to 853]

OUTCOME MEASURES:

1. Primary Outcome: Reactive Hyperemia Index (RHI) by Peripheral Arterial Tonometry (PAT)
Description: Ratio of the average pulse wave amplitude (PWA) over a 1 minute interval starting 1 minute following cuff release to the pre-occlusion PWA (average over 3.5 minutes pre-cuff inflation)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 45 | 41
ratio | 1.98 [1.79 to 2.48] | 2.15 [1.71 to 2.58]

2. Secondary Outcome: Soluble Biomarkers (Fasting Lipid Panel, hsCRP, IL-6, D-dimer, sICAM-1, sE-selectin, Lp-PLA2, sCD14, sCD163)
Description: Serum hsCRP
Time Frame: Baseline
Population: All participants with available data.
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Group A (HIV/HCV Coinfected): HIV+/HCV viremic
- Group B (HIV Monoinfected): HIV+/HCV-
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 35 | 41
mg/L | 0.6 [0.2 to 2.1] | 1.3 [0.8 to 2.8]

3. Secondary Outcome: Reactive Hyperemia Index (RHI)
Description: as for outcome 1
Time Frame: Week 52
Measure: Median (Inter-Quartile Range); unit: ratio
Groups:
- Group A (HIV/HCV Coinfected): HIV+/HCV+, HCV treated
- Group B (HIV Monoinfected): HIV+/HCV- at study entry
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 31 | 29
ratio | 1.88 [1.65 to 2.55] | 2.09 [1.64 to 2.42]

4. Secondary Outcome: Soluble Biomarkers (Fasting Lipid Panel, hsCRP, IL-6, D-dimer, sICAM-1, sE-selectin, Lp-PLA2, sCD14, sCD163)
Description: Serum hsCRP
Time Frame: Week 52
Population: All participants with available data.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 30 | 16
mg/L | 1.05 [0.40 to 2.50] | 1.0 [0.75 to 1.40]

5. Secondary Outcome: Insulin Resistance by HOMA-IR
Description: fasting insulin (μU/mL) x fasting glucose (mg/dl) / 405
Time Frame: Baseline
Population: All participants with available data.
Measure: Median (Inter-Quartile Range); unit: HOMA-IR score
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 35 | 41
HOMA-IR score | 3.86 [1.70 to 5.40] | 2.24 [1.36 to 3.17]

6. Secondary Outcome: Insulin Resistance by HOMA-IR
Description: fasting insulin (μU/mL) x fasting glucose (mg/dl) / 405
Time Frame: Week 52
Population: All participants with available data
Measure: Median (Inter-Quartile Range); unit: HOMA-IR score
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 30 | 16
HOMA-IR score | 2.77 [2.06 to 4.72] | 2.13 [1.33 to 4.78]

7. Secondary Outcome: Framingham Risk Score (FRS), 10-year Risk (%)
Description: Estimate of 10-year risk for developing coronary heart disease (CHD), calculated as described in ATP III Executive Summary, JAMA, May 16, 2001-Vol 285, No. 19. Range of values is <1 to >/= 30% Higher risk % is worse predicted outcome.
Time Frame: Baseline
Population: All participants with available data
Measure: Median (Inter-Quartile Range); unit: percent, 10-year risk
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 45 | 41
percent, 10-year risk | 6.0 [2.0 to 8.0] | 6.0 [3.0 to 10.0]

8. Secondary Outcome: Framingham Risk Score (FRS), 10-year Risk (%)
Description: as for outcome 7
Time Frame: Week 52
Population: All participants with available data
Measure: Median (Inter-Quartile Range); unit: percent, 10-year risk
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 30 | 16
percent, 10-year risk | 6.0 [4.0 to 8.0] | 5.0 [1.0 to 8.0]

9. Secondary Outcome: Change in RHI
Time Frame: Baseline to Week 52
Population: All with available data
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 31 | 29
ratio | -0.16 [-0.43 to -0.06] | -0.03 [-0.32 to 0.05]

10. Secondary Outcome: Change in Level of Each Soluble Biomarker (Components of Fasting Lipid Panel, hsCRP, IL-6, D-dimer, sICAM-1, sE-selectin, Lp-PLA2, sCD14, sCD163)
Description: Change in serum hsCRP level
Time Frame: Baseline to Week 52
Population: All participants with available data
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Group A (HIV/HCV Coinfected): HIV+/HCV viremic, HCV treated
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 27 | 16
mg/L | 0.40 [0.00 to 1.20] | 0.00 [-0.45 to 0.45]

11. Secondary Outcome: Change in HOMA-IR
Time Frame: Baseline to Week 52
Population: All participants with available data
Measure: Median (Inter-Quartile Range); unit: HOMA-IR score
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 27 | 16
HOMA-IR score | 0.34 [-1.23 to 1.66] | 0.28 [-0.59 to 1.82]

12. Secondary Outcome: Change in Framingham Risk Score (10-year Risk, %)
Description: Change in estimated 10-year risk (% risk) for developing coronary heart disease (CHD). Positive value indicates increase in estimated 10-year risk for CHD from baseline to Week 52. Negative value indicates decrease in estimated 10-year risk for CHD from baseline to Week 52.
Time Frame: Baseline to Week 52
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
Number analyzed (Participants) | 27 | 16
percent | 1.0 [0.0 to 2.0] | 0 [-1.0 to 0.5]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Group A (HIV/HCV Coinfected) | Group B (HIV Monoinfected)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT02597790/Prot_SAP_000.pdf